CLINICAL TRIAL: NCT00179465
Title: Addition of Tiagabine to Second-Generation Antipsychotics in the Treatment of Recent-Onset Schizophrenia by Modification of Developmental Reorganization of the Prefrontal Cortex
Brief Title: Treating Schizophrenia by Correcting Abnormal Brain Development
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Tsung-Ung Wilson Woo, Assistant Professor of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004P000078
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia
Keywords: Treatment; fMRI; Cognition; Brain development
MeSH Terms: conditions — Schizophrenia | interventions — Tiagabine; Antipsychotic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antipsychotic plus study drug (Active Comparator): Half of the subjects will receive the study medications in addition to their ongoing antipsychotic regimen.
  Interventions: Drug: Tiagabine
- Antipsychotics plus placebo (Placebo Comparator): Half of the subjects will receive placebo in addition to their antipsychotic regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiagabine — Up to 36 mg daily
  Other Names: Antipsychotic
  Arms: Antipsychotic plus study drug
Drug: Placebo — Placebo
  Other Names: Antipsychotic
  Arms: Antipsychotics plus placebo

SUMMARY:
The purpose of this study is to determine whether treatment with tiagabine (Gabitril) during the early course of schizophrenia can fundamentally correct the brain deficits associated with the disease.

This study is funded by the National Institutes of Health.

DETAILED DESCRIPTION:
It is hypothesized that enhancement of GABA neurotransmission during the early course of the illness by tiagabine (Gabitril), a GABA transporter GAT-1-specific inhibitor and a FDA-approved anticonvulsant, will improve both clinical symptoms and working memory in schizophrenia. This improvement is postulated to be the result of tiagabine-mediated modification of the developmental synaptic pruning of prefrontal cortical circuitry. The occurrence of circuitry modification after tiagabine treatment will be assessed by the following independent methodologic approaches: MRI morphometric analysis of prefrontal gray matter volume and fMRI measurements of brain activity patterns during performance of tasks that probe working memory.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for the diagnosis of schizophrenia, with onset of psychotic symptoms within the past 3 years.
* Currently on second-generation antipsychotics for at least 3 months.
* Age 18-25, otherwise healthy.

Exclusion Criteria:

* Diagnosis of schizoaffective disorder.
* Has failed two or more clinically adequate antipsychotic trials.
* History of seizures or any neurologic disorders.
* Pregnant or nursing women.
* Known HIV infection.
* Actively suicidal.
* History of any substance dependence.
* Currently meets criteria for substance abuse/dependence.
* Other MRI exclusion criteria per Radiology Department protocols.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2003-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Functions-Working Memory | Working memory will be assessed at baseline and at 6-month time point to see if working memory changes after 6 months compared to baseline measurement
  Working memory will be assessed using the n-back working memory test
Neurocognitive Functions-Executive Function | Executive function will be assessed at baseline and at 6-month time point to see if executive function changes after 6 months compared to baseline measure
  Executive function, which is a complex form of working memory, will be assessed using the MATRICS (Measurement and Treatment Research to Improve Cognition in Schizophrenia) battery

SECONDARY OUTCOMES:
Clinical symptoms | Symptoms will be assessed at baseline and at 6-month time point to see if symptoms change after 6 months compared to baseline measures
  Positive and negative symptoms will be quantified using PANSS (positive and negative symptom scale)

CONTACTS AND LOCATIONS:
Overall Officials: T.-U. Wilson Woo, M.D., Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Woo TU, Crowell AL. Targeting synapses and myelin in the prevention of schizophrenia. Schizophr Res. 2005 Mar 1;73(2-3):193-207. doi: 10.1016/j.schres.2004.07.022. PMID 15653262
- [Background] Woo TU, Whitehead RE, Melchitzky DS, Lewis DA. A subclass of prefrontal gamma-aminobutyric acid axon terminals are selectively altered in schizophrenia. Proc Natl Acad Sci U S A. 1998 Apr 28;95(9):5341-6. doi: 10.1073/pnas.95.9.5341. PMID 9560277
- [Background] Woo TU, Spencer K, McCarley RW. Gamma oscillation deficits and the onset and early progression of schizophrenia. Harv Rev Psychiatry. 2010 May-Jun;18(3):173-89. doi: 10.3109/10673221003747609. PMID 20415633